CLINICAL TRIAL: NCT03073486
Title: A Randomized, Double-blind, Vehicle Controlled, Efficacy and Safety Study of Olumacostat Glasaretil Gel in Subjects With Acne Vulgaris
Brief Title: A Study of Olumacostat Glasaretil Gel in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRM01B-ACN04
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Results first posted 2019-02-05 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olumacostat Glasaretil Gel, 5.0% (Experimental): Olumacostat Glasaretil Gel, 5.0%, applied twice daily to the face for 12 weeks
  Interventions: Drug: Olumacostat Glasaretil Gel, 5.0%
- Olumacostat Glasaretil Gel, Vehicle (Placebo Comparator): Olumacostat Glasaretil Gel, Vehicle, applied twice daily to the face for 12 weeks
  Interventions: Other: Olumacostat Glasaretil Gel, Vehicle

INTERVENTIONS:
Drug: Olumacostat Glasaretil Gel, 5.0% — Gel containing Olumacostat Glasaretil
  Other Names: DRM01
  Arms: Olumacostat Glasaretil Gel, 5.0%
Other: Olumacostat Glasaretil Gel, Vehicle — Vehicle (placebo) gel
  Arms: Olumacostat Glasaretil Gel, Vehicle

SUMMARY:
The objectives of this study are to assess the safety and efficacy of Olumacostat Glasaretil Gel compared to vehicle in patients with acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and, for subjects under legal adult age, signed assent
* Age ≥ 9 years
* Clinical diagnosis of facial acne vulgaris defined as:

  * At least 20 inflammatory lesions, and
  * At least 20 non-inflammatory lesions, and
  * Investigator Global Assessment of 3 or greater

Exclusion Criteria:

* Active cystic acne or acne conglobata, acne fulminans, and secondary acne
* Two or more active nodulocystic lesions on the face
* Clinically significant abnormal laboratory or ECG result
* Subjects who are actively participating in an experimental therapy study or who have received experimental therapy within 30 days or 5 half-lives (whichever is longer) of the Baseline visit
* Treatment with over-the-counter topical medications for the treatment of acne vulgaris including benzoyl peroxide, topical anti-inflammatory medications, corticosteroids, α-hydroxy/glycolic acid on the face within 2 weeks prior to Baseline
* Treatment with systemic antibiotics or systemic anti-acne drugs or topical retinoid within 4 weeks prior to Baseline
* Treatment with a new hormonal therapy or dose change to existing hormonal therapy within 12 weeks prior to Baseline (hormonal therapies include, but are not limited to, estrogenic and progestational agents such as birth control pills).
* Use of androgen receptor blockers (such as spironolactone or flutamide) within 2 weeks prior to Baseline.
* Oral retinoid use (e.g., isotretinoin) within 12 months prior to Baseline or vitamin A supplements greater than 10,000 units/day within 6 months prior to Baseline
* Facial procedures (chemical or laser peel, microdermabrasion, etc.) within the past 8 weeks

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Zib, Study Director — Dermira, Inc.
Locations (46):
- United States (36):
  - Avant Research Associates, LLC, Guntersville, Alabama
  - Advanced Research Associates, Glendale, Arizona
  - Dermatology Trial Associates, Bryant, Arkansas
  - Northwest Arkansas Clinical Trials Center, Rogers, Arkansas
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Advanced Skincare Surgery & MedCenter, Fullerton, California
  - Northern California Research, Sacramento, California
  - TCR Medical Corporation, San Diego, California
  - Radiant Research, Inc., Santa Rosa, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Center for Clincial and Cosmetic Research, Aventura, Florida
  - Florida Academic Centers Research & Education, Coral Gables, Florida
  - Aby's New GEneration Research Inc., Hialeah, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Floridian Research Institute, Miami, Florida
  - Pioneer Clinical Research, Pembroke Pines, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - MOORE Clinical Research, Inc, Tampa, Florida
  - Visions Clinical Research, Wellington, Florida
  - Marietta Dermatology Clinical Research, Inc., Marietta, Georgia
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Henry Ford Medical Center, New Center One, Detroit, Michigan
  - JDR Dermatology Research, LLC, Las Vegas, Nevada
  - Skin Search of Rochester, Inc., Rochester, New York
  - Sterling Research Group, Cincinnati, Ohio
  - The Skin Wellness Center, Knoxville, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Avant Research Associates, Beaumont, Texas
  - Synexus US, LP, dba, Research Across America, Dallas, Texas
  - Suzanne Bruce and Associates, P.A. The Center for Skin, Houston, Texas
  - Austin Institute for Clinical Research, Inc, Pflugerville, Texas
  - Houston Center for Clinical Research, Sugar Land, Texas
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
  - Premier Clinical Research, Spokane, Washington
- Australia (5):
  - The Skin Centre, Benowa
  - Premier Specialists, Kogarah
  - Sinclair Dermatology, Melbourne
  - Burswood Dermatology, Victoria Park
  - Veracity Clinical Research, Woolloongabba
- Canada (5):
  - Enverus Medical Research, Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - DermEdge Research, Mississauga, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - XLR8 Medical Research, Windsor, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olumacostat Glasaretil Gel, 5.0% | Olumacostat Glasaretil Gel, Vehicle
Started | 493 | 251
Completed | 405 | 207
Not Completed | 88 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olumacostat Glasaretil Gel, 5.0% | Olumacostat Glasaretil Gel, Vehicle | Total
Number analyzed (Participants) | 493 | 251 | 744
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 304 | 147 | 451
  Between 18 and 65 years | 189 | 104 | 293
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.2 (6.98) | 19.2 (7.26) | 19.2 (7.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 294 | 145 | 439
  Male | 199 | 106 | 305
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 88 | 52 | 140
  Not Hispanic or Latino | 393 | 196 | 589
  Unknown or Not Reported | 12 | 3 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 35 | 9 | 44
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 90 | 54 | 144
  White | 342 | 178 | 520
  More than one race | 21 | 9 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 44 | 22 | 66
  United States | 393 | 200 | 593
  Australia | 56 | 29 | 85
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Type is a scale to numerically classify skin color, defined by the response to ultraviolet (UV) light with the following categories:
  Type I Burns easily, rarely tans Type II Burns easily, tans minimally Type III Burns moderately, tans gradually Type IV Burns minimally, tans well Type V Rarely burns, tans profusely Type VI Never burns, deeply pigmented
  Participants
    Type I | 33 | 13 | 46
    Type II | 99 | 61 | 160
    Type III | 133 | 58 | 191
    Type IV | 112 | 57 | 169
    Type V | 51 | 26 | 77
    Type VI | 65 | 36 | 101

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Change in Acne Lesion Counts (Inflammatory) From Baseline to Week 12
Description: Mean absolute change in acne lesion counts (inflammatory) from baseline to Week 12
Time Frame: Baseline and Week 12
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Deviation); unit: Lesions
Arm/Group | Olumacostat Glasaretil Gel, 5.0% | Olumacostat Glasaretil Gel, Vehicle
Number analyzed (Participants) | 493 | 251
Lesions | -17.0 (12.16) | -15.4 (11.95)
Statistical Analysis 1: Comparison: Olumacostat Glasaretil Gel, 5.0% vs Olumacostat Glasaretil Gel, Vehicle; Test type: Other; p = 0.2301, ANCOVA; Ranked ANCOVA, Markov Chain Monte Carlo (MCMC) Multiple Imputation

2. Primary Outcome: Mean Absolute Change in Acne Lesion Counts (Non-inflammatory) From Baseline to Week 12
Description: Mean absolute change in acne lesion counts (non-inflammatory) from baseline to Week 12
Time Frame: Baseline and Week 12
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Deviation); unit: Lesions
Arm/Group | Olumacostat Glasaretil Gel, 5.0% | Olumacostat Glasaretil Gel, Vehicle
Number analyzed (Participants) | 493 | 251
Lesions | -18.0 (23.37) | -17.6 (22.64)
Statistical Analysis 1: Comparison: Olumacostat Glasaretil Gel, 5.0% vs Olumacostat Glasaretil Gel, Vehicle; Test type: Other; p = 0.6888, ANCOVA; Ranked ANCOVA, Markov Chain Monte Carlo (MCMC) Multiple Imputation

3. Primary Outcome: Percentage of Subjects Who Achieved ≥ 2-grade Improvement and a Grade of 0 or 1 in the Investigator Global Assessment of Acne (IGA) From Baseline to Week 12
Description: Percentage of subjects who achieved ≥ 2-grade improvement and a grade of 0 or 1 in the investigator global assessment of acne (IGA) from baseline to Week 12
  Scoring Criteria for Investigator Global Assessment 0 - Clear skin with no inflammatory or noninflammatory lesions
  1. - Almost clear; rare noninflammatory lesions with no more than one small inflammatory lesion
  2. - Mild severity; greater than Grade 1; some noninflammatory lesions with no more than a few inflammatory lesions (papules/pustules only, no nodular lesions)
  3. - Moderate severity; greater than Grade 2; up to many noninflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesion
  4. - Severe; greater than Grade 3; up to many noninflammatory and inflammatory lesions, but no more than a few nodular lesions
Time Frame: Baseline and Week 12
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Olumacostat Glasaretil Gel, 5.0% | Olumacostat Glasaretil Gel, Vehicle
Number analyzed (Participants) | 493 | 251
Participants
  Success | 80 | 30
  Failure | 413 | 221
Statistical Analysis 1: Comparison: Olumacostat Glasaretil Gel, 5.0% vs Olumacostat Glasaretil Gel, Vehicle; Test type: Other; p = 0.1361, Regression, Logistic; Logistic Regression (Firth's Penalized Likelihood), MCMC Multiple Imputation

ADVERSE EVENTS:
Time Frame: Baseline to Week 12
Description: The Total Participants at risk are based on the Safety Population defined as Participants who were randomized and received at least one confirmed dose of study drug.
Arm/Group | Olumacostat Glasaretil Gel, 5.0% | Olumacostat Glasaretil Gel, Vehicle
All-Cause Mortality (participants affected / at risk) | 0/491 | 0/248
Serious Adverse Events (participants affected / at risk) | 1/491 | 0/248
Other Adverse Events (participants affected / at risk) | 108/491 | 28/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olumacostat Glasaretil Gel, 5.0% (N=491) | Olumacostat Glasaretil Gel, Vehicle (N=248)
Suicidal ideation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olumacostat Glasaretil Gel, 5.0% (N=491) | Olumacostat Glasaretil Gel, Vehicle (N=248)
Application site dryness (General disorders) | 15 | 2
Application site erythema (General disorders) | 28 | 3
Application site pain (General disorders) | 30 | 6
Application site pruritus (General disorders) | 38 | 17
Nasopharyngitis (Infections and infestations) | 9 | 7
Upper respiratory tract infection (Infections and infestations) | 20 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT03073486/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT03073486/SAP_001.pdf